CLINICAL TRIAL: NCT00493051
Title: A Randomized, Double-Blind, Placebo-Controlled, Single- and Double-Dose, Comparator Arm (Standard of Care), Multicenter Phase 2b Study of Topical GAM501 (Ad5PDGF-B/Bovine Type I Collagen Gel) in the Treatment of Non-Healing Diabetic Ulcers of the Lower Extremities
Brief Title: Phase 2b Study of GAM501 in the Treatment of Diabetic Ulcers of the Lower Extremities
Acronym: MATRIX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tissue Repair Company (Industry)
Collaborators: Cardium Therapeutics (Industry)
Responsible Party: Barbara Sosnowski/ Chief Operating Officer, Tissue Repair Company
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SWHI-03
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Diabetic Foot
Keywords: diabetes; nonhealing; ulcers; neuropathic
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Ulcer | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Other): Standardized Wound Care
  Interventions: Other: Standard of care
- 2 (Placebo Comparator): Placebo 1 dose
  Interventions: Biological: Placebo
- 3 (Placebo Comparator): Placebo 2 doses
  Interventions: Biological: Placebo
- 4 (Active Comparator): Active 1 dose
  Interventions: Biological: GAM501
- 5 (Active Comparator): Active 2 doses
  Interventions: Biological: GAM501

INTERVENTIONS:
Biological: GAM501 — Ad5PDGF-B formulated in a collagen gel
  Other Names: Excellarate
  Arms: 4; 5
Biological: Placebo — Collagen gel
  Arms: 2; 3
Other: Standard of care — moist dressing changes daily
  Arms: 1

SUMMARY:
This is a Phase 2b, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of one or two applications of topically applied GAM501 (Ad5PDGF-B/Bovine Type I Collagen Gel) in subjects ≥ 18 years old with non-healing diabetic foot ulcers. Approximately 210 adult subjects with Type I or Type II diabetes mellitus will be enrolled at approximately 30 investigational sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of diabetes mellitus (Type I or II) requiring insulin or hypoglycemic agents to control blood sugars.
* Cutaneous, lower extremity ulcer of the foot that is ≥1.5 and ≤10.0 cm² in size and Wagner Classification Grade 1 in appearance. Note - Ulcer area must be calculated at Screening Visit and on the Treatment Day (Day 1) using measurements obtained by tracing the ulcer perimeter after debridement to confirm patient eligibility prior to randomization.
* Documented ulcer presence for ≥6 weeks prior to signing the informed consent form
* Recently debrided ulcer (within 2 weeks from screening visit)
* Ulcer free of all necrotic soft tissue
* Affected limb transcutaneous partial pressure oxygen (TcpO2) >40mmHg; or a toe pressure ≥40mmHg; or a Doppler waveform consistent with adequate flow in the foot (biphasic or triphasic waveforms) at screening
* Inability to perceive 10 grams pressure using a Semmes-Weinstein 5.07 monofilament in the peri-ulcer area
* Willing to adhere to wearing off-loading orthopedic shoe for up to 16 weeks (i.e., through 2 weeks after ulcer closure) starting on Day -14 (the first day of the screening run-in period)
* Willing to adhere to wearing customized shoes during the durability phase of the study
* Females of child-bearing potential must have a negative serum beta human chorionic gonadotropin hormone (ßhCG) test result from a sample obtained in the 7 days prior to Treatment Day 1 and be neither breastfeeding nor intending to become pregnant during the study
* All individuals (study patients/partners) of childbearing potential must agree to use a method of contraception deemed acceptable by the Investigator or agree to remain abstinent throughout the study
* Be able to understand and sign an informed consent form before entering into the study, and must be willing to comply with all study procedures

Exclusion Criteria:

* Any unstable medical condition judged by the Investigator or Medical Monitor that would cause the study to be detrimental to the patient
* Hemoglobin Alc (HbA1c) test result of >12% documented at the Screening Visit
* Ulcers caused primarily by untreated vascular insufficiency; or ulcers with an etiology not related to diabetes
* Ulcers on the heel
* More than three ulcers on the target lower extremity
* The ulcer to be studied is not anatomically distinct from another ulcer(s) (i.e., separated by <1 cm from another ulcer or would interfere with standard of care treatment of another ulcer). Only a single ulcer can be treated in this study.
* Ulcers which decrease in area by >30% during the screening 2-week run-in period
* Ulcers with underlying osteomyelitis
* Patients presenting with the clinical characteristics of cellulitis at the ulcer site (suppurative inflammation involving particularly the subcutaneous tissue, often mild erythema, tenderness, malaise, chills and fever)
* If either beta hemolytic streptococci (in any amount) or total bacterial load of >1e6 CFU/gram of tissue is present in the screening biopsy sample at the ulcer site, the patient should be given a single 7-day course of topical antibiotics and then redebrided and biopsied for quantitative culture. A second biopsy exceeding the limits above will result in exclusion from the study due to the high risk of local infection than may adversely affect ulcer closure.
* Revascularization surgery on the leg with the wound to be treated ≤8 weeks prior to signing the informed consent form
* Surgery to lengthen Achilles tendon on the leg with the wound to be treated ≤8 weeks prior to signing the informed consent form
* Necrosis, purulence, or sinus tracts that cannot be removed by debridement on foot to be treated
* Needs concurrent topical antimicrobials to treat the ulcer site, or received such therapies within 7 days prior to signing the informed consent form
* Received dermal substitute or living skin equivalent (e.g., Dermagraft® or Appligraf®) within 30 days prior to signing the informed consent form
* Received prior PDGF-BB (Regranex®/becaplermin) therapy within 30 days prior to signing the informed consent form
* Has known sensitivity to products of bovine origin
* Life expectancy of less than 12 months
* Patients with a definite diagnosis of any immunodeficiency disorder
* Viral hepatitis [patient must have a negative hepatitis B surface-antigen (HBsAg) and hepatitis C antibody (HepCAb) test results obtained within 2 weeks prior to the Treatment Day (Day 1)]
* Active, uncontrolled connective tissue disease
* Renal failure as defined by serum creatinine >2.5 mg/dL
* Liver function studies (e.g., AST, ALT) that are >2.0 times upper limit of normal
* Poor nutritional status as measured by serum albumin <3.0 g/dL
* Active cancer or a history of cancer in the 5 years prior to signing the informed consent form (however, history of basal cell carcinoma is allowed)
* Active (i.e., recent onset of erythema, edema, and increased temperature of the foot with normal radiographs ) Charcot or other structural deformity that would prevent adequate off-loading of the study foot
* Treatment with any systemic corticosteroid, immunosuppressive chemotherapeutic agent, antiviral, or previous/current radiation therapy to lower extremity within 30 days prior to signing the informed consent form
* Received another investigational drug or biologic within 30 days prior to signing the informed consent form or currently participating in an investigational drug or biologic study
* A psychiatric condition or chronic alcohol or drug abuse problem, determined from the patient's medical history, which in the Investigator's opinion may pose a threat to patient compliance
* History of non-compliance with treatment or clinical visit attendance (i.e., this study requires that patients will comply with the protocol and ulcer care regimen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Effect of GAM501 on the incidence of complete ulcer closure | Week 12 or earlier

SECONDARY OUTCOMES:
Time to complete ulcer closure | The time from treatment start to first visit when ulcer closure is documented
The absolute change and percent change in ulcer area | From baseline ulcer area and measured at weekly intervals through week 12
The durability of ulcer closure | Measured at 4 week intervals for 12 weeks from date of ulcer closure
Ulcer healing trajectories will be assessed by plots of percentage of ulcer closure versus time | Week 12 or earlier
Safety and tolerance | Week 12 or earlier

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Kittrelle, MD, Study Chair — Tissue Repair Company, 6740 Top Gun St, San Diego, CA 92121 USA, 858-259-4511
Locations (29):
- United States (29):
  - Baptist Medical Center South, Montgomery, Alabama
  - Banner Baywood Medical Center, Mesa, Arizona
  - Associated Foot & Ankle Specialists, Phoenix, Arizona
  - Aung Foothealth Clinics, Tuscon, Arizona
  - Absolute Foot Care, Chula Vista, California
  - Dr. Roy Kroeker DPM, Fresno, California
  - Dr. Jagpreet Mukker, Fresno, California
  - Long Beach VA Health Care System, Long Beach, California
  - LAC-USC Medical Center, Los Angeles, California
  - Innovative Medical Technologies, Los Angeles, California
  - UCLA Medical Center Olive View, Sylmar, California
  - Foot Doctors of Watsonville, Watsonville, California
  - North American Center for Limb Preservation, New Haven, Connecticut
  - Providence Hospital Clinical Research Center, Washington D.C., District of Columbia
  - Bay Pines VAHCS, Bay Pines, Florida
  - Karr Foot Kare, Lakeland, Florida
  - University of Miami, Miami, Florida
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - Division of Wound Healing & Regenerative Medicine NYU School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Leigh Valley Hospital, Allentown, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Warren General Hospital, Warren, Pennsylvania
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - St. Joseph Medical Center, Houston, Texas
  - South Texas Foot Institute, San Antonio, Texas

REFERENCES:
- [Background] Steed DL, Attinger C, Colaizzi T, Crossland M, Franz M, Harkless L, Johnson A, Moosa H, Robson M, Serena T, Sheehan P, Veves A, Wiersma-Bryant L. Guidelines for the treatment of diabetic ulcers. Wound Repair Regen. 2006 Nov-Dec;14(6):680-92. doi: 10.1111/j.1524-475X.2006.00176.x. No abstract available. PMID 17199833
- See also: American Diabetes Association Web Page — http://www.diabetes.org/
- See also: MATRIX Phase 2b study website — http://www.diabeticfootstudy.com